CLINICAL TRIAL: NCT01909570
Title: Randomized Clinical Trial Comparing Elective Single Embryo Transfer Plus Single Embryo Cryotransfer vs Double Embryo Transfer
Brief Title: eSET Plus Single Embryo Cryotransfer vs Double Embryo Transfer
Acronym: eSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Ana Clavero Gilabert, PhD MD, University Hospital Virgen de las Nieves
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FIS09/1968
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Infertility; Pregnancy, Multiple
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elective single embryo transfer (Experimental): After the FIV/ICSI procedure, in this arm the embryo transfer would be of a single embryo followed by the cryotransfer or a single embryo in case of no fresh conception
  Interventions: Procedure: Elective single embryo transfer
- Double embryo transfer (Active Comparator): After the FIV/ICSI procedure, in this arm the embryo transfer woub be of two fresh embryos
  Interventions: Procedure: Double embryo transfer

INTERVENTIONS:
Procedure: Elective single embryo transfer — After the FIV/ICSI procedure, the embryo transfer in this arm would be of one embryo followed by the cryotransfer of one embryo in case of no conception in the fresh cycle.
  Arms: Elective single embryo transfer
Procedure: Double embryo transfer — After the FIV/ICSI procedure, the embryo transfer in this arm would be of two fresh embryos
  Arms: Double embryo transfer

SUMMARY:
The purpose of this study is to determine whether a policy of elective single embryo transfer (eSET) plus single embryo cryotransfer is as effective as a double embryo transfer in terms of clinical pregnancy rate

DETAILED DESCRIPTION:
The objective is to evaluate the In Vitro Fertilization/Intracytoplasmic Sperm Inyection (IVF/ICSI) results in terms of clinical pregnancy and multiple pregnancy rates, comparing elective single embryo transfer plus cryotransfer of one embryo if pregnancy is not achieved, with double embryo transfer.

This is a prospective randomized study, including couples arriving to the Reproductive Unit of the Hospital Universitario Virgen de las Nieves. All these patients had good reproductive prognosis and had been asigned randomly to one of the following groups: Group 1: elective single embryo transfer. In the case pregnancy is not achieved a cryotransfer of one embryo will be carried out. Group 2: elective double embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* women less tan 38 years
* women Body Mass Index (BMI) between 19-39 kg/m2
* Follicle-Stimulating Hormone (FSH) <15 mUI/mL on cycle third day
* First IVF/ICSI cycle or second after a positive pregnancy test in the first one

Exclusion Criteria:

* More tan five years of infertility
* Previous uterus surgery
* Uterus malformations
* More tan one miscarriage

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Clavero, PhD, Principal Investigator — Investigator and laboratory specialist
Locations (1):
- Unidad de gestión clínica de ginecología y obstetricia. Instituto Biosanitario de Granada.Hospital Universitario Virgen de las Nieves, Granada, Spain

REFERENCES:
- [Derived] Lopez-Regalado ML, Clavero A, Gonzalvo MC, Serrano M, Martinez L, Mozas J, Rodriguez-Serrano F, Fontes J, Castilla JA. Randomised clinical trial comparing elective single-embryo transfer followed by single-embryo cryotransfer versus double embryo transfer. Eur J Obstet Gynecol Reprod Biol. 2014 Jul;178:192-8. doi: 10.1016/j.ejogrb.2014.04.009. Epub 2014 Apr 19. PMID 24798072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from January 2010 to December 2012. The location of the recruitment was University Hospital of Virgen de las Nieves in Granada.
Pre-assignment Details: A total of 194 women aged under 38 years were included in the study. Of these, 19 women were not randomised. The reasons were refusion to participate (n= 6), economic reasons (n = 2), participating in another study (n= 7) and not meeting criteria in further evaluation (n = 4).
Groups:
- Elective Single Embryo Transfer: Elective single embryo transfer plus single embryo cryotransfer in case of no fresh conception
- Double Embryo Transfer: Transfer of two fresh embryos
Period: Overall Study
Arm/Group | Elective Single Embryo Transfer | Double Embryo Transfer
Started | 84 | 91
Completed | 57 | 64
Not Completed | 27 | 27

BASELINE CHARACTERISTICS:
Population: Women aged under 38 years, with BMI between 19-29 kg/m2, FSH <15mUI/mL on the third day and first cycle of IVF/ICSI or second cycle after a prior attempt with a positive pregnancy test result. The infertile period must be less of five years, without previous uterine surgery, uterine malformations, neither repeated spontaneous abortions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elective Single Embryo Transfer | Double Embryo Transfer | Total
Number analyzed (Participants) | 84 | 91 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (3.6) | 31.7 (3.8) | 32.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 91 | 175
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 84 | 91 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 84 | 91 | 175

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate
Description: A clinical pregnancy was defined by the presence of a gestational sac with heartbeat on transvaginal ultrasonography at the 7th weeks of pregnancy
Time Frame: Seven weeks after embryo transfer
Population: as for baseline characteristics
Measure: Number; unit: percentage of pregnancy per transfer
Arm/Group | Elective Single Embryo Transfer | Double Embryo Transfer
Number analyzed (Participants) | 84 | 91
percentage of pregnancy per transfer | 44.0 | 37.4

2. Secondary Outcome: Multiple Pregnancy Rate
Description: A multiple clinical pregnancy was defined by the presence of more than one gestational sac with heartbeat on transvaginal ultrasonography at the 7th weeks of pregnancy
Time Frame: Seven weeks after embryo transfer
Population: as for baseline characteristics
Measure: Number; unit: percentage of multiple pregnancies
Arm/Group | Elective Single Embryo Transfer | Double Embryo Transfer
Number analyzed (Participants) | 84 | 91
percentage of multiple pregnancies | 0 | 26.4

3. Other Pre Specified Outcome: Live Birth Delivery Rate
Description: The delivery of a healthy child (o two)
Time Frame: 38 weeks after embryo transfer
Population: as for baseline characteristics
Measure: Number; unit: percentage of live birth
Arm/Group | Elective Single Embryo Transfer | Double Embryo Transfer
Number analyzed (Participants) | 84 | 91
percentage of live birth | 45.2 | 41.8

ADVERSE EVENTS:
Arm/Group | Elective Single Embryo Transfer | Double Embryo Transfer
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/91
Other Adverse Events (participants affected / at risk) | 3/84 | 5/91
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elective Single Embryo Transfer (N=84) | Double Embryo Transfer (N=91)
premature birth (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) — Child birth before 37 gestational weeks
Hiperstimulation Ovarian Syndrome (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Syndrome of hiperactivation of ovarian function due to fertility treatments

LIMITATIONS AND CAVEATS:
Our study could have been complemented by improved embryo selection, using a time-lapse system.

Another limitation of our study is that after devitrification, blastocyst culture was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No